CLINICAL TRIAL: NCT04872842
Title: Establishment of Online Registration Platform for Unruptured Intracranial Aneurysms Based on 100 Regional Medical Centers in China and Population Follow-up Study
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Peking University Third Hospital (Other); Beijing Sanbo Brain Hospital (Other); Beijing Chao Yang Hospital (Other); Binzhou Renmin Hospital (Unknown); Fujian Medical University Union Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); Guangzhou Red Cross Hospital (Other); The First Affiliated Hospital of Haerbin Medical University (Unknown); The Affiliated Hospital of Qingdao University (Other); Shanxi Provincial People's Hospital (Other Government); Beijing Tsinghua Changgeng Hospital (Other); RenJi Hospital (Other); Sichuan Provincial People's Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Affiliated Hospital of Kunming Medical University (Unknown); Beijing Unimed Technology Company (Unknown)
Responsible Party: Principal Investigator, Wang Shuo, Director of Department of Cerebrovascular Neurosurgery, Beijing Tiantan Hospital
Other Study IDs: 82071296
Record Dates: First submitted 2021-04-22; First posted 2021-05-05 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Intracranial Aneurysm
Keywords: intracranial aneurysm; online registration platform; artificial intelligence; multidimensional model
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- unstable intracranial aneurysms: Unstable intracranial aneurysms are defined as the intracranial aneurysms that grows or ruptures.
  Interventions: Other: Obervation
- stable intracranial aneurysms: Stable intracranial aneurysms are defined as the intracranial aneurysms that have no significant morphological changes.
  Interventions: Other: Obervation

INTERVENTIONS:
Other: Obervation — This study is an observational study without any intervention

SUMMARY:
In this study, 20 regional neurosurgery centers across the country will be included, and the study cohort will be constructed on the basis of the IARP-CP cohort.The artificial intelligence platform was used to analyze the clinical, morphological, hemodynamics, aneurysm wall characteristics and other factors of unruptured aneurysms, as well as the relationship between these factors and the risk of aneurysm instability, seek the potential risk factors, and finally establish a multi-dimensional prediction model of rupture risk of intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old;
2. At least one unruptured intracranial aneurysm was found by CTA;
3. No relevant symptoms, receiving non-operative and conservative observation treatment;
4. Signing the informed consent.

Exclusion Criteria:

1. Other cerebrovascular structural lesions (such as cerebrovascular malformation and arteriovenous fistula) or craniocerebral tumors;
2. Fusiform or dissecting aneurysms;
3. Traumatic, mycotic and atrial myxoma associated aneurysms;
4. Suffering from systemic connective tissue diseases, such as polycystic kidney disease;
5. Expectant survival of no more than 3 years due to other diseases or poor general conditions;
6. Patients refuse to follow up or cannot communicate with them due to mental diseases;
7. Pregnant women or participating in other aneurysm related studies.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Aneurysm rupture | 2 years

SECONDARY OUTCOMES:
Aneurysm growth | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Wang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Liu Q, Li J, Zhang Y, Leng X, Mossa-Basha M, Levitt MR, Wang S, Zhu C. Association of calcium channel blockers with lower incidence of intracranial aneurysm rupture and growth in hypertensive patients. J Neurosurg. 2023 Jan 27;139(3):651-660. doi: 10.3171/2022.12.JNS222428. Print 2023 Sep 1. PMID 36708539